CLINICAL TRIAL: NCT00889941
Title: Effect of Preoperative Pupil Size on Quality of Vision After Wavefront-Guided LASIK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Edward Manche, MD, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-02082009-1758
Record Dates: First submitted 2009-02-12; First posted 2009-04-29 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- small (Active Comparator)
  Interventions: Procedure: LASIK
- medium (Active Comparator)
  Interventions: Procedure: LASIK
- large (Active Comparator)
  Interventions: Procedure: LASIK

INTERVENTIONS:
Procedure: LASIK — laser-assisted in situ keratomileusis
  Other Names: laser-assisted in situ keratomileusis

SUMMARY:
The purpose of this study is to evaluate whether the size of the pupil has an effect on quality of vision in patients undergoing LASIK surgery.

DETAILED DESCRIPTION:
Purpose: To prospectively evaluate the effect of preoperative pupil size on quality of vision after wavefront-guided LASIK.

Methods: Fifty-one patients underwent LASIK for low myopia and completed questionnaires regarding specific visual symptoms before and after surgery. Each eye was evaluated postoperatively at 1-week, 1-, 3-, 6- and 12-months. Pupils were stratified according to size: small (<5.5mm), medium (5.5 to 6.0mm) and large (>6.0mm). Mesopic pupil size and preoperative and postoperative variables were evaluated using analysis of variance (ANOVA). A regression model was also performed to determine the correlation between mean spherical equivalent and cylinder and visual symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. no more than 6.00 D of spherical myopia
2. no more than 3.00 D of refractive astigmatism
3. a stable refraction (less than 0.50D per year of sphere or cylinder)
4. a corneal diameter of less than 11.0 mm to allow for suction ring fixation
5. discontinuation of soft contact wear at least 7 days prior to preoperative evaluation
6. visual acuity correctable to at least 20/20
7. age older than 21 years
8. ability to participate in follow-up examinations for 12 months after LASIK surgery

Exclusion Criteria:

1. use of rigid gas permeable contact lens
2. severe dry eye symptoms
3. severe blepharitis
4. anterior segment abnormalities (i.e. cataracts, corneal scarring, or neovascularization within 1 mm of intended ablation zone)
5. recurrent corneal erosion
6. severe basement membrane disease
7. progressive or unstable myopia or keratoconus
8. unstable corneal mires on central keratometry
9. corneal thickness in which LASIK procedure would result in less than 250 microns of remaining posterior corneal thickness below the flap postoperatively
10. baseline standard manifest refraction of more than 0.75 D in sphere power
11. or a difference of greater than 0.50 D in cylinder power compared with baseline standard cycloplegic refraction
12. a baseline standard cycloplegic refraction differing more than 0.75 in sphere, 0.50 D in cylinder
13. have a different type of astigmatism (i.e. with-the-rule) when the cylinder is greater than 0.50D compared to baseline standard cycloplegic refraction
14. preoperative assessment of ocular topography and/or aberrations indicates that either eye is not suitable candidate for LASIK vision correction procedure (i.e. forme fruste keratoconus
15. corneal warpage, or pellucid marginal degeneration)
16. previous intraocular or corneal surgery
17. history of herpes zoster or simplex keratitis
18. patients on systemic corticosteroid or immunosuppressive therapy
19. immunocompromised subjects or clinically significant atopic disease
20. connective tissue disease
21. diabetes
22. steroid responder
23. macular pathology
24. pregnant or lactating patients
25. patients with sensitivity to planned study concomitant medications
26. patients participating in another ophthalmic drug or device clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2004-05; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annie Chan, Sub-Investigator — Stanford University; Edward E. Manche, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States